CLINICAL TRIAL: NCT01559441
Title: The Effects of Beetroot Juice on Postprandial Vascular Activity After a High-fat Meal in Overweight and Slightly Obese Men
Brief Title: Beetroot Juice and Postprandial Vascular Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: METC 11-3-085
Record Dates: First submitted 2012-03-12; First posted 2012-03-21 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Dyslipidemia
Keywords: beetroot juice; nitrate; vascular activity; postprandial state
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beetroot juice (Experimental)
  Interventions: Dietary Supplement: Beetroot Juice with oral fat load
- Carbohydrate control drink (Placebo Comparator)
  Interventions: Dietary Supplement: Carbohydrate control drink with oral fat load

INTERVENTIONS:
Dietary Supplement: Beetroot Juice with oral fat load — 140mL (9.6 mmol nitrate) beetroot juice (Beet It, James White drinks Ltd)
  Arms: Beetroot juice
Dietary Supplement: Carbohydrate control drink with oral fat load — 140 mL (low-nitrate) carbohydrate control drink
  Arms: Carbohydrate control drink

SUMMARY:
Increased postprandial lipemia may increase the risk for cardiovascular diseases. An important mechanistic link between lipemia following a high-fat meal and adverse cardiovascular events is lipid-mediated endothelial activation. Therefore, it is important to identify nutrients that can neutralize this acute vascular disturbance.

The investigators hypothesize that beetroot juice, a food rich in inorganic nitrate, could improve vascular activity during the postprandial phase.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years
* Quetelet-index between 28-35 kg/m2
* Mean serum triacylglycerol ≤1.7 mmol/L
* No indication for treatment with cholesterol-lowering drugs according to the Dutch Cholesterol Consensus
* No current smoker
* No diabetic patients or individuals receiving antidiabetic medication
* No familial hypercholesterolemia
* No abuse of drugs
* Less than 21 alcoholic consumptions per week
* Stable body weight (weight gain or loss <3 kg in the past three months)
* No use of medication known to affect serum lipid metabolism
* No severe medical conditions that might interfere with the study, such as high blood pressure, epilepsy, asthma, allergies, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* No active cardiovascular disease like congestive heart failure or recent (<6 months) event (acute myocardial infarction, cerebro vascular accident)
* Willingness to stop the consumption of foods rich in nitrates 3 weeks before the start of the study. Vegetables such as beets, celery, radishes, turnips and spinach are rich in nitrates
* Willingness to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visits

Exclusion Criteria:

* Women
* Quetelet-index between <28 or >35 kg/m2
* Mean serum triacylglycerol ≥1.7 mmol/L
* Indication for treatment with cholesterol-lowering drugs according to the Dutch Cholesterol Consensus
* Current smoker
* Diabetic patients or individuals receiving antidiabetic medication
* Familial hypercholesterolemia
* Abuse of drugs
* More than 21 alcoholic consumptions per week
* Unstable body weight (weight gain or loss >3 kg in the past three months)
* Use of use of medication known to affect serum lipid metabolism
* No severe medical conditions that might interfere with the study, such as high blood pressure, epilepsy, asthma, allergies, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or recent (<6 months) event (acute myocardial infarction, cerebro vascular accident)
* Use of an investigational product within the previous 1 month
* Not willing to stop the consumption of foods rich in nitrates 3 weeks before the start of the study
* Not willing to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study, during the study or for 4 weeks after completion of the study
* Not or difficult to venipuncture as evidenced during the screening visits

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Vascular activity | Change from baseline at 2 hours after meal consumption
  Flow-mediated dilation (FMD) of the brachial artery

SECONDARY OUTCOMES:
Arterial stiffness | Change from baseline at 3 hours after meal consumption
  Pulse wave analysis (PWA) and velocity (PWV)
Microcirculatory effects | Change from baseline at 3 hours after meal consumption
  Retinal imaging
Metabolic risk markers related to the metabolic syndrome | During 4 hours after meal consumption
  Changes in biomarkers for low-grade systemic inflammation and endothelial activation.
Postprandial lipid metabolism | During 4 hours after meal consumption
Postprandial glucose metabolism | During 4 hours after meal consumption

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P Mensink, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands